CLINICAL TRIAL: NCT02853890
Title: " 7 Days Survey of Obstetric Analgesia/Anesthesia in France" (EPIDOL)
Brief Title: Management of Obstetrical Pain: " 7 Days Survey of Obstetric Analgesia/Anesthesia in France"
Acronym: Epidol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0047
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Birth
Keywords: Birth; obstetric analgesia; obstetric anesthesia
MeSH Terms: interventions — Parturition

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pregnant woman
  Interventions: Other: Questionnaires during hospitalization for delivery

INTERVENTIONS:
Other: Questionnaires during hospitalization for delivery — Questionnaires during hospitalization for delivery (one questionnaire completed by doctors about different technic of analgesia and anesthesia and one questionnaire completed by women about pain, and feeling about the different techniques of analgesia and anesthesia used during delivery, eventually caesarean section or uterine revision)

SUMMARY:
Obstetric analgesia is a requirement of our times. The different applicable methods vary in effectiveness. The essential part is represented by epidural analgesia which remains one of the most effective methods. It is important to know other methods to respond to all requests. The applications of these methods, patient satisfaction and psychic experience, complications or incidents remain poorly or partially evaluated in France.

The main objective is to describe the different techniques of anesthesia/analgesia actually used in France for the management of pain during vaginal deliveries and cesarean sections on a representative sample of all maternity hospitals at a given time(7 days per maternity hospital, 63 maternity hospitals (levels I,II,III), so about 2500 births).

Secondary objectives will be multiple :

* Describe the results of analgesic methods on the physical pain of patients during labor by a global visual analog scale
* Describe the feeling of pregnant women relative to the different anesthesic and analgesic techniques, by an analysis of the questionnaire responses
* Describe the frequency of adverse events of birth

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in a maternity hospital for delivery during the 7 days defined for the study will be included

Exclusion Criteria:

* Patients under 18 years old
* Lack of understanding of the French language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All woman patients hospitalized for delivery
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Type of analgesia techniques | Day 0
  description of the different techniques of analgesia during labor, uterine revision and eventually cesarean section assessed by a questionnaire
Type of anesthesia techniques | Day 0
  description of the different techniques of anesthesia during labor, uterine revision and eventually cesarean section assessed by a questionnaire

SECONDARY OUTCOMES:
physical pain assessed by using a visual analog scale. | Day 1
Assessment of the feeling of pregnant women about the analgesic and anesthesic techniques by a questionnaire | Day 2
Collect of adverse events | Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Chassard, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chassard D, Langlois-Jacques C, Naaim M, Galetti S, Bouvet L, Coz E, Ecochard R, Portefaix A, Kassai-Koupai B; CARO Group. Anesthesia practices for management of labor pain and cesarean delivery in France (EPIDOL): A cross-sectional survey. Anaesth Crit Care Pain Med. 2023 Dec;42(6):101302. doi: 10.1016/j.accpm.2023.101302. Epub 2023 Sep 12. PMID 37709198